CLINICAL TRIAL: NCT00296270
Title: "Myths and Facts" About the Flu: Health Education Campaigns Can Reduce Vaccination Intentions
Brief Title: Memory for Flu Facts and Myths and Effects on Vaccine Intentions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: RIR13914
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2006-02-24 (Estimated); Status verified 2006-02

CONDITIONS: Influenza Vaccines
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Behavioral: Memory for truth

SUMMARY:
Objectives: To determine whether people systematically misremember the "myths" (false information) as true, and to assess effects on perceptions of risk and behavioral intentions.

DETAILED DESCRIPTION:
Public information campaigns often warn people about false and unreliable medical claims by juxtaposing "myths" and "facts." The effectiveness of such communications has rarely been assessed. We assessed whether people systematically misremember the "myths" (false information) as true, and to assess effects on perceptions of risk and behavioral intentions.

In an experimental study, participants read either a published CDC flyer on "Facts and Myths" about the flu vaccine, or a "Facts Only" version; a separate control group read no flyer. Participants completed the outcome measures either immediately or after 30 minutes.

Primary measures were memory for information about the flu presented in the flyer, ratings of perceived risks associated with the flu, and personal intentions to get vaccinated in the upcoming season.

After a delay of 30 minutes, participants who read the "Facts and Myths" flyer systematically misremembered myths as facts. Both versions of the flyer had the immediate effect of increasing intentions to get a flu vaccine, compared to the control group. After 30 minutes, however, participants who read the "Facts and Myths" flyer reported lower intentions to get vaccinated, compared to those who read the same flyer with no delay, and compared to all participants who read the "Facts Only" flyer.

In sum, people show a bias to think that incompletely remembered information is true, turning "myths" into "facts." Hence public information campaigns should emphasize information that is true. Repeating false information, even as a warning, can create the unintended consequence of belief in the information.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to read and write fluent English

Exclusion Criteria:

-

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175
Dates: Start 2005-03; Study Completion 2005-06

PRIMARY OUTCOMES:
Memory for truth of information in a flyer.

SECONDARY OUTCOMES:
Intention to get flu vaccine in upcoming season.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Skurnik, PhD, Principal Investigator — Rotman School of Management, University of Toronto
Locations (2):
- University of Michigan, Ann Arbor, Michigan, United States
- Rotman School of Management, University of Toronto, Toronto, Ontario, Canada